CLINICAL TRIAL: NCT03499600
Title: Improving Satisfaction, Engagement and Clinical Outcomes Among Traditionally Underserved Children Through Cultural Formulation
Brief Title: Improving Satisfaction, Engagement and Outcomes Among Traditionally Underserved Children Through Cultural Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: University of Miami (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 106618; R36MH116677-01 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Disruptive Behavior
Keywords: Cultural assessment; Engagement; Diverse Populations
MeSH Terms: conditions — Problem Behavior | interventions — chemotactic factor inactivator

STUDY DESIGN:
Intervention Model Description: Randomized control trial in which participants are randomly assigned to either receive a diagnostic and clinical assessment plus the cultural formulation interview (CA and CFI) or the diagnostic and clinical assessment (CA).
Who Masked: Participant, Outcomes Assessor
Masking Description: Coders assessing therapist fidelity to the CFI are kept unaware of the condition to which each participant is assigned. Participants will also be unaware of the condition to which they have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Assessment and CFI (Experimental): CA and CFI families will receive the Cultural Formulation Interview prior to their standard Clinical Assessment during their intake.
  Interventions: Behavioral: Clinical Assessment and CFI
- Clinical Assessment Only (Active Comparator): CA families will receive a standard Clinical Assessment during intake.
  Interventions: Behavioral: Clinical Assessment

INTERVENTIONS:
Behavioral: Clinical Assessment and CFI — CA and CFI families will participate in the Cultural Formulation Interview prior to their standard intake.
  Arms: Clinical Assessment and CFI
Behavioral: Clinical Assessment — CA families will participate their standard intake procedures.
  Arms: Clinical Assessment Only

SUMMARY:
The project at the center of this proposal will leverage a pilot randomized design to examine initial feasibility and preliminary effects of augmenting usual mental health evaluation procedures with a structured person-centered assessment tool that specifically considers the cultural context of patient mental health problems (i.e., the Cultural Formulation Interview; CFI) on parent satisfaction, engagement and clinical child outcomes in the treatment of early child behavior problems. Additional analyses will explore whether traditional barriers (e.g., stigma, ethnic identity, and daily stress) moderate the effects of the CFI on satisfaction, engagement and treatment outcomes.

DETAILED DESCRIPTION:
This project is leveraging a pilot randomized design to evaluate initial feasibility and preliminarily examine whether augmenting assessment procedures for child behavior problems with the CFI improves satisfaction with assessment procedures and treatment, parent engagement in subsequent behavior parent training, and ultimately clinical child outcomes. Exploratory analyses will further consider whether traditional barriers to care moderate outcomes. The study is being conducted within a large South Florida mental health network serving predominately low-income minority families obtaining parent training for early child behavior problems. Participating families will be randomized at baseline to receive either the standard diagnostic and clinical assessment (CA) or CA+CFI.

Specifically, the investigators are interested in assessing study feasibility. Feasibility of recruitment and randomization, study retention, and condition integrity will be monitored. Additionally, clinician reports of CFI feasibility, acceptability and clinical utility will be examined. An additional main outcome will be initial satisfaction directly after the interview. It is hypothesized that families in the CA+CFI group will report higher levels of initial satisfaction than the CA group. A secondary goal is to assess preliminary effects of administering the CFI on treatment satisfaction, engagement and clinical child outcomes. Parents and therapists will report on their satisfaction with treatment. Engagement outcomes will be measured via: (a) initial session attendance, (b) drop out rate (c) session attendance rate, (d) homework completion rate, and (e) therapeutic alliance. Clinical outcomes will be measured via parent ratings of child behavior problems and parent time to skill mastery. It is hypothesized that CA+CFI families will demonstrate improved satisfaction, engagement and clinical outcomes relative to CA families. Further exploratory analyses will examine individual differences in effects related to traditional barriers to care. Exploratory analyses will examine stigma, ethnic identity, and daily stress as moderators of the effects of CFI administration on satisfaction, engagement and clinical outcomes. It is hypothesized that CFI effects will be particularly strong for families who experience greater traditional barriers to care.

ELIGIBILITY:
Inclusion Criteria:

* Child with elevated behavior problems
* Child is between ages 2-7 years (inclusive)
* Family seeking services at one of the University of Miami PCIT-Community Connect Centers

Exclusion Criteria:

* Parent is actively abusing illegal substances
* Child is younger than 2 years of age
* Child is older than 7 years of age

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Mailman Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will use a controlled access approach, using a robust system to review requests and provide secure access to de-identified data

REFERENCES:
- [Background] Aggarwal NK. Cultural formulations in child and adolescent psychiatry. J Am Acad Child Adolesc Psychiatry. 2010 Apr;49(4):306-9. No abstract available. PMID 20410723
- [Background] Aggarwal NK, Desilva R, Nicasio AV, Boiler M, Lewis-Fernandez R. Does the Cultural Formulation Interview for the fifth revision of the diagnostic and statistical manual of mental disorders (DSM-5) affect medical communication? A qualitative exploratory study from the New York site. Ethn Health. 2015;20(1):1-28. doi: 10.1080/13557858.2013.857762. Epub 2013 Nov 15. PMID 25372242
- [Background] Aggarwal NK, Glass A, Tirado A, Boiler M, Nicasio A, Alegria M, Wall M, Lewis-Fernandez R. The development of the DSM-5 Cultural Formulation Interview-Fidelity Instrument (CFI-FI): a pilot study. J Health Care Poor Underserved. 2014 Aug;25(3):1397-417. doi: 10.1353/hpu.2014.0132. PMID 25130248
- [Background] Aggarwal NK, Lam P, Castillo EG, Weiss MG, Diaz E, Alarcon RD, van Dijk R, Rohlof H, Ndetei DM, Scalco M, Aguilar-Gaxiola S, Bassiri K, Deshpande S, Groen S, Jadhav S, Kirmayer LJ, Paralikar V, Westermeyer J, Santos F, Vega-Dienstmaier J, Anez L, Boiler M, Nicasio AV, Lewis-Fernandez R. How Do Clinicians Prefer Cultural Competence Training? Findings from the DSM-5 Cultural Formulation Interview Field Trial. Acad Psychiatry. 2016 Aug;40(4):584-91. doi: 10.1007/s40596-015-0429-3. Epub 2015 Oct 8. PMID 26449983
- [Background] Aggarwal NK, Nicasio AV, DeSilva R, Boiler M, Lewis-Fernandez R. Barriers to implementing the DSM-5 cultural formulation interview: a qualitative study. Cult Med Psychiatry. 2013 Sep;37(3):505-33. doi: 10.1007/s11013-013-9325-z. PMID 23836098
- [Background] Akincigil A, Olfson M, Siegel M, Zurlo KA, Walkup JT, Crystal S. Racial and ethnic disparities in depression care in community-dwelling elderly in the United States. Am J Public Health. 2012 Feb;102(2):319-28. doi: 10.2105/AJPH.2011.300349. Epub 2011 Dec 15. PMID 22390446
- [Background] Alegría, M., Green, J. G., McLaughlin, K. A., & Loder, S. (2015). Disparities in child and adolescent mental health and mental health services in the US.
- [Background] Alegria M, Vallas M, Pumariega AJ. Racial and ethnic disparities in pediatric mental health. Child Adolesc Psychiatr Clin N Am. 2010 Oct;19(4):759-74. doi: 10.1016/j.chc.2010.07.001. PMID 21056345
- [Background] American Psychiatric Association (2000). Diagnostic and statisticalmanual of mental disorders (4th ed., text rev.). Washington, DC: Author.
- [Background] American Psychiatric Association (2013). Diagnostic and statistical manual of mental disorders (5th ed.). Arlington, VA: American Psychiatric Publishing.
- [Background] Barkley RA, Shelton TL, Crosswait C, Moorehouse M, Fletcher K, Barrett S, Jenkins L, Metevia L. Multi-method psycho-educational intervention for preschool children with disruptive behavior: preliminary results at post-treatment. J Child Psychol Psychiatry. 2000 Mar;41(3):319-32. PMID 10784079
- [Background] Blanco C, Patel SR, Liu L, Jiang H, Lewis-Fernandez R, Schmidt AB, Liebowitz MR, Olfson M. National trends in ethnic disparities in mental health care. Med Care. 2007 Nov;45(11):1012-9. doi: 10.1097/MLR.0b013e3180ca95d3. PMID 18049340
- [Background] Briggs-Gowan MJ, Carter AS, Skuban EM, Horwitz SM. Prevalence of social-emotional and behavioral problems in a community sample of 1- and 2-year-old children. J Am Acad Child Adolesc Psychiatry. 2001 Jul;40(7):811-9. doi: 10.1097/00004583-200107000-00016. PMID 11437020
- [Background] Burke JD, Waldman I, Lahey BB. Predictive validity of childhood oppositional defiant disorder and conduct disorder: implications for the DSM-V. J Abnorm Psychol. 2010 Nov;119(4):739-51. doi: 10.1037/a0019708. PMID 20853919
- [Background] Burnett-Zeigler I, Lee Y, Bohnert KM. Ethnic Identity, Acculturation, and 12-Month Psychiatric Service Utilization Among Black and Hispanic Adults in the U.S. J Behav Health Serv Res. 2018 Jan;45(1):13-30. doi: 10.1007/s11414-017-9557-8. PMID 28492979
- [Background] Bussing R, Zima BT, Gary FA, Garvan CW. Barriers to detection, help-seeking, and service use for children with ADHD symptoms. J Behav Health Serv Res. 2003 Apr-Jun;30(2):176-89. doi: 10.1007/BF02289806. PMID 12710371
- [Background] Bussing R, Zima BT, Perwien AR, Belin TR, Widawski M. Children in special education programs: attention deficit hyperactivity disorder, use of services, and unmet needs. Am J Public Health. 1998 Jun;88(6):880-6. doi: 10.2105/ajph.88.6.880. PMID 9618613
- [Background] Butler AM, Titus C. Systematic Review of Engagement in Culturally Adapted Parent Training for Disruptive Behavior. J Early Interv. 2015 Dec;37(4):300-318. doi: 10.1177/1053815115620210. PMID 27429537
- [Background] Chronis AM, Jones HA, Raggi VL. Evidence-based psychosocial treatments for children and adolescents with attention-deficit/hyperactivity disorder. Clin Psychol Rev. 2006 Aug;26(4):486-502. doi: 10.1016/j.cpr.2006.01.002. Epub 2006 Feb 17. PMID 16483703
- [Background] Cunningham CE, Boyle M, Offord D, Racine Y, Hundert J, Secord M, McDonald J. Tri-ministry study: correlates of school-based parenting course utilization. J Consult Clin Psychol. 2000 Oct;68(5):928-33. PMID 11068980
- [Background] Eiraldi RB, Mazzuca LB, Clarke AT, Power TJ. Service Utilization among ethnic minority children with ADHD: a model of help-seeking behavior. Adm Policy Ment Health. 2006 Sep;33(5):607-22. doi: 10.1007/s10488-006-0063-1. PMID 16862391
- [Background] Eyberg SM, Nelson MM, Boggs SR. Evidence-based psychosocial treatments for children and adolescents with disruptive behavior. J Clin Child Adolesc Psychol. 2008 Jan;37(1):215-37. doi: 10.1080/15374410701820117. PMID 18444059
- [Background] Eyberg, S. M., & Pincus, D. (1999). ECBI & SESBI-R: Eyberg child behavior inventory and Sutter-Eyberg student behavior inventory-revised: Professional manual. Psychological Assessment Resources
- [Background] Fabrega H Jr, Ulrich R, Mezzich JE. Do Caucasian and black adolescents differ at psychiatric intake? J Am Acad Child Adolesc Psychiatry. 1993 Mar;32(2):407-13. doi: 10.1097/00004583-199303000-00023. PMID 8444771
- [Background] Fantuzzo, J., Stoltzfus, J., Lutz, M. N., Hamlet, H., Balraj, V., Turner, C., & Mosca, S. (1999). An evaluation of the special needs referral process for low-income preschool children with emotional and behavioral problems. Early Childhood Research Quarterly, 14(4), 465-482
- [Background] Fernandez, M. (2011). Treatment outcome for low socioeconomic status African American families in parent child interaction therapy: A pilot study. Child and Family Behavior Therapy, 33, 32-48.
- [Background] Forehand R, Kotchick BA. Cultural Diversity: A Wake-Up Call for Parent Training - Republished Article. Behav Ther. 2016 Nov;47(6):981-992. doi: 10.1016/j.beth.2016.11.010. Epub 2016 Nov 10. PMID 27993345
- [Background] Flores G; Committee On Pediatric Research. Technical report--racial and ethnic disparities in the health and health care of children. Pediatrics. 2010 Apr;125(4):e979-e1020. doi: 10.1542/peds.2010-0188. Epub 2010 Mar 29. PMID 20351000
- [Background] Garland AF, Lau AS, Yeh M, McCabe KM, Hough RL, Landsverk JA. Racial and ethnic differences in utilization of mental health services among high-risk youths. Am J Psychiatry. 2005 Jul;162(7):1336-43. doi: 10.1176/appi.ajp.162.7.1336. PMID 15994717
- [Background] Gopalan G, Goldstein L, Klingenstein K, Sicher C, Blake C, McKay MM. Engaging families into child mental health treatment: updates and special considerations. J Can Acad Child Adolesc Psychiatry. 2010 Aug;19(3):182-96. PMID 20842273
- [Background] Gross DA, Belcher HM, Ofonedu ME, Breitenstein S, Frick KD, Chakra B. Study protocol for a comparative effectiveness trial of two parent training programs in a fee-for-service mental health clinic: can we improve mental health services to low-income families? Trials. 2014 Mar 1;15:70. doi: 10.1186/1745-6215-15-70. PMID 24581245
- [Background] Hall, LA. Social support, everyday stressors, and maternal mental health (Unpublished doctoral dissertation). Chapel Hill, NC: University of North Carolina; 1983.
- [Background] Hall GC, Ibaraki AY, Huang ER, Marti CN, Stice E. A Meta-Analysis of Cultural Adaptations of Psychological Interventions. Behav Ther. 2016 Nov;47(6):993-1014. doi: 10.1016/j.beth.2016.09.005. Epub 2016 Sep 30. PMID 27993346
- [Background] Hatcher, R. L., & Gillaspy, J. A. (2006). Development and validation of a revised short version of the Working Alliance Inventory. Psychotherapy Research, 16(1), 12-25.
- [Background] Herschell, A. D., Calzada, E. J., Eyberg, S. M., & McNeil, C. B. (2002). Parent-child interaction therapy: New directions in research. Cognitive and Behavioral Practice, 9(1), 9-16.
- [Background] Hoza B. Peer functioning in children with ADHD. J Pediatr Psychol. 2007 Jul;32(6):655-63. doi: 10.1093/jpepsy/jsm024. Epub 2007 Jun 7. PMID 17556400
- [Background] Ingoldsby EM. Review of Interventions to Improve Family Engagement and Retention in Parent and Child Mental Health Programs. J Child Fam Stud. 2010 Oct 1;19(5):629-645. doi: 10.1007/s10826-009-9350-2. PMID 20823946
- [Background] Kataoka SH, Zhang L, Wells KB. Unmet need for mental health care among U.S. children: variation by ethnicity and insurance status. Am J Psychiatry. 2002 Sep;159(9):1548-55. doi: 10.1176/appi.ajp.159.9.1548. PMID 12202276
- [Background] Kazdin, A. E., Mazurick, J. L., & Bass, D. (1993). Risk for attrition in treatment of antisocial children and families. Journal of Clinical Child Psychology, 22(1), 2-16.
- [Background] Kazdin AE, Whitley M, Marciano PL. Child-therapist and parent-therapist alliance and therapeutic change in the treatment of children referred for oppositional, aggressive, and antisocial behavior. J Child Psychol Psychiatry. 2006 May;47(5):436-45. doi: 10.1111/j.1469-7610.2005.01475.x. PMID 16671927
- [Background] Kim-Cohen J, Caspi A, Moffitt TE, Harrington H, Milne BJ, Poulton R. Prior juvenile diagnoses in adults with mental disorder: developmental follow-back of a prospective-longitudinal cohort. Arch Gen Psychiatry. 2003 Jul;60(7):709-17. doi: 10.1001/archpsyc.60.7.709. PMID 12860775
- [Background] Kirmayer LJ. Beyond the 'new cross-cultural psychiatry': cultural biology, discursive psychology and the ironies of globalization. Transcult Psychiatry. 2006 Mar;43(1):126-44. doi: 10.1177/1363461506061761. PMID 16671396
- [Background] Kirmayer, L. J., Rousseau, C., Rosenberg, E., Clarke, H., Saucier, J. F., Sterlin, C., ... & Latimer, E. (2001). Development and evaluation of a cultural consultation service in mental health. Culture and Mental Health Research Unit, Report, 11.
- [Background] Lau, A. S. (2006). Making the case for selective and directed cultural adaptations of evidence-based treatments: examples from parent training. Clinical psychology: Science and Practice, 13(4), 295-310.
- [Background] Lavigne JV, Lebailly SA, Gouze KR, Binns HJ, Keller J, Pate L. Predictors and correlates of completing behavioral parent training for the treatment of oppositional defiant disorder in pediatric primary care. Behav Ther. 2010 Jun;41(2):198-211. doi: 10.1016/j.beth.2009.02.006. Epub 2009 Dec 5. PMID 20412885
- [Background] Leijten P, Raaijmakers MA, de Castro BO, Matthys W. Does socioeconomic status matter? A meta-analysis on parent training effectiveness for disruptive child behavior. J Clin Child Adolesc Psychol. 2013;42(3):384-92. doi: 10.1080/15374416.2013.769169. Epub 2013 Mar 5. PMID 23461526
- [Background] Lewis-Fernandez R, Aggarwal NK, Baarnhielm S, Rohlof H, Kirmayer LJ, Weiss MG, Jadhav S, Hinton L, Alarcon RD, Bhugra D, Groen S, van Dijk R, Qureshi A, Collazos F, Rousseau C, Caballero L, Ramos M, Lu F. Culture and psychiatric evaluation: operationalizing cultural formulation for DSM-5. Psychiatry. 2014 Summer;77(2):130-54. doi: 10.1521/psyc.2014.77.2.130. PMID 24865197
- [Background] Lewis-Fernandez R, Aggarwal NK, Lam PC, Galfalvy H, Weiss MG, Kirmayer LJ, Paralikar V, Deshpande SN, Diaz E, Nicasio AV, Boiler M, Alarcon RD, Rohlof H, Groen S, van Dijk RC, Jadhav S, Sarmukaddam S, Ndetei D, Scalco MZ, Bassiri K, Aguilar-Gaxiola S, Ton H, Westermeyer J, Vega-Dienstmaier JM. Feasibility, acceptability and clinical utility of the Cultural Formulation Interview: mixed-methods results from the DSM-5 international field trial. Br J Psychiatry. 2017 Apr;210(4):290-297. doi: 10.1192/bjp.bp.116.193862. Epub 2017 Jan 19. PMID 28104738
- [Background] Lewis-Fernandez R, Balan IC, Patel SR, Sanchez-Lacay JA, Alfonso C, Gorritz M, Blanco C, Schmidt A, Jiang H, Schneier F, Moyers TB. Impact of motivational pharmacotherapy on treatment retention among depressed Latinos. Psychiatry. 2013 Fall;76(3):210-22. doi: 10.1521/psyc.2013.76.3.210. PMID 23965261
- [Background] Lewis-Fernández, R., Aggarwal, N. K., Hinton, L., Hinton, D. E., & Kirmayer L. .J., (Eds.). (2015). DSM-5® handbook on the cultural formulation interview. American Psychiatric Association Publishing.
- [Background] Matos M, Bauermeister JJ, Bernal G. Parent-child interaction therapy for Puerto Rican preschool children with ADHD and behavior problems: a pilot efficacy study. Fam Process. 2009 Jun;48(2):232-52. doi: 10.1111/j.1545-5300.2009.01279.x. PMID 19579907
- [Background] Matos M, Torres R, Santiago R, Jurado M, Rodriguez I. Adaptation of parent-child interaction therapy for Puerto Rican families: a preliminary study. Fam Process. 2006 Jun;45(2):205-22. doi: 10.1111/j.1545-5300.2006.00091.x. PMID 16768019
- [Background] McCabe K, Yeh M. Parent-child interaction therapy for Mexican Americans: a randomized clinical trial. J Clin Child Adolesc Psychol. 2009 Sep;38(5):753-9. doi: 10.1080/15374410903103544. PMID 20183659
- [Background] McKay MM, Pennington J, Lynn CJ, McCadam K. Understanding urban child mental health l service use: two studies of child, family, and environmental correlates. J Behav Health Serv Res. 2001 Nov;28(4):475-83. doi: 10.1007/BF02287777. PMID 11732249
- [Background] McKay MM, Bannon WM Jr. Engaging families in child mental health services. Child Adolesc Psychiatr Clin N Am. 2004 Oct;13(4):905-21, vii. doi: 10.1016/j.chc.2004.04.001. PMID 15380788
- [Background] McKay MM, McCadam K, Gonzales JJ. Addressing the barriers to mental health services for inner city children and their caretakers. Community Ment Health J. 1996 Aug;32(4):353-61. doi: 10.1007/BF02249453. PMID 8840078
- [Background] McMahon RJ, Frick PJ. Evidence-based assessment of conduct problems in children and adolescents. J Clin Child Adolesc Psychol. 2005 Sep;34(3):477-505. doi: 10.1207/s15374424jccp3403_6. PMID 16026215
- [Background] Miranda J, Bernal G, Lau A, Kohn L, Hwang WC, LaFromboise T. State of the science on psychosocial interventions for ethnic minorities. Annu Rev Clin Psychol. 2005;1:113-42. doi: 10.1146/annurev.clinpsy.1.102803.143822. No abstract available. PMID 17716084
- [Background] Merikangas KR, He JP, Burstein M, Swendsen J, Avenevoli S, Case B, Georgiades K, Heaton L, Swanson S, Olfson M. Service utilization for lifetime mental disorders in U.S. adolescents: results of the National Comorbidity Survey-Adolescent Supplement (NCS-A). J Am Acad Child Adolesc Psychiatry. 2011 Jan;50(1):32-45. doi: 10.1016/j.jaac.2010.10.006. Epub 2010 Dec 3. PMID 21156268
- [Background] Mezzich JE, Caracci G, Fabrega H Jr, Kirmayer LJ. Cultural formulation guidelines. Transcult Psychiatry. 2009 Sep;46(3):383-405. doi: 10.1177/1363461509342942. PMID 19837778
- [Background] National Institute of Mental Health. Blueprint for change: research on child and adolescent mental health. Rockville: US Department of Health and Human Services Administration, Center of Mental Health Services, National Institute of Health, National Institute of Mental Health; 2001.
- [Background] Nixon RD, Sweeney L, Erickson DB, Touyz SW. Parent-child interaction therapy: one- and two-year follow-up of standard and abbreviated treatments for oppositional preschoolers. J Abnorm Child Psychol. 2004 Jun;32(3):263-71. doi: 10.1023/b:jacp.0000026140.60558.05. PMID 15228175
- [Background] Nock MK, Kazdin AE, Hiripi E, Kessler RC. Lifetime prevalence, correlates, and persistence of oppositional defiant disorder: results from the National Comorbidity Survey Replication. J Child Psychol Psychiatry. 2007 Jul;48(7):703-13. doi: 10.1111/j.1469-7610.2007.01733.x. PMID 17593151
- [Background] Novins DK, Bechtold DW, Sack WH, Thompson J, Carter DR, Manson SM. The DSM-IV Outline for Cultural Formulation: a critical demonstration with American Indian children. J Am Acad Child Adolesc Psychiatry. 1997 Sep;36(9):1244-51. doi: 10.1097/00004583-199709000-00017. PMID 9291726
- [Background] Owens J. Early Childhood Behavior Problems and the Gender Gap in Educational Attainment in the United States. Sociol Educ. 2016;89(3):236-258. doi: 10.1177/0038040716650926. Epub 2016 Jun 22. PMID 30393398
- [Background] Phinney, J. S., & Ong, A. D. (2007). Conceptualization and measurement of ethnic identity: Current status and future directions. Journal of Counseling Psychology, 54(3), 271.
- [Background] Qi, C. H., & Kaiser, A. P. (2003). Behavior problems of preschool children from low-income families review of the literature. Topics in Early Childhood Special Education, 23(4), 188-216.
- [Background] Richardson LA. Seeking and obtaining mental health services: what do parents expect? Arch Psychiatr Nurs. 2001 Oct;15(5):223-31. doi: 10.1053/apnu.2001.27019. PMID 11584351
- [Background] Rowe R, Costello EJ, Angold A, Copeland WE, Maughan B. Developmental pathways in oppositional defiant disorder and conduct disorder. J Abnorm Psychol. 2010 Nov;119(4):726-38. doi: 10.1037/a0020798. PMID 21090876
- [Background] Schim SM, Doorenbos AZ, Miller J, Benkert R. Development of a Cultural Competence Assessment instrument. J Nurs Meas. 2003 Spring-Summer;11(1):29-40. doi: 10.1891/jnum.11.1.29.52062. PMID 15132010
- [Background] Spoth, R., Redmond, C., Hockaday, C., & Shin, C. Y. (1996). Barriers to participation in family skills preventive interventions and their evaluations: A replication and extension. Family Relations, 247-254.
- [Background] Sue S, Fujino DC, Hu LT, Takeuchi DT, Zane NW. Community mental health services for ethnic minority groups: a test of the cultural responsiveness hypothesis. J Consult Clin Psychol. 1991 Aug;59(4):533-40. doi: 10.1037//0022-006x.59.4.533. PMID 1918557
- [Background] Sue S, Zane N. The role of culture and cultural techniques in psychotherapy. A critique and reformulation. Am Psychol. 1987 Jan;42(1):37-45. doi: 10.1037//0003-066x.42.1.37. No abstract available. PMID 3565913
- [Background] Takeuchi J. Treatment of a biracial child with schizophreniform disorder: cultural formulation. Cultur Divers Ethnic Minor Psychol. 2000 Feb;6(1):93-101. doi: 10.1037/1099-9809.6.1.93. PMID 10975171
- [Background] Turner EA. The parental attitudes toward psychological services inventory: adaptation and development of an attitude scale. Community Ment Health J. 2012 Aug;48(4):436-49. doi: 10.1007/s10597-011-9432-7. Epub 2011 Jun 21. PMID 21691821
- [Background] Yasui M, Hipwell AE, Stepp SD, Keenan K. Psychocultural Correlates of Mental Health Service Utilization Among African American and European American Girls. Adm Policy Ment Health. 2015 Nov;42(6):756-66. doi: 10.1007/s10488-014-0610-0. PMID 25380787
- [Background] Young AS, Rabiner D. Racial/ethnic differences in parent-reported barriers to accessing children's health services. Psychol Serv. 2015 Aug;12(3):267-73. doi: 10.1037/a0038701. Epub 2015 Jan 19. PMID 25602502
- [Derived] Sanchez AL, Jent J, Aggarwal NK, Chavira D, Coxe S, Garcia D, La Roche M, Comer JS. Person-Centered Cultural Assessment Can Improve Child Mental Health Service Engagement and Outcomes. J Clin Child Adolesc Psychol. 2022 Jan-Feb;51(1):1-22. doi: 10.1080/15374416.2021.1981340. Epub 2021 Dec 14. PMID 34905434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families were recruited and randomized from August 2017 to October 2018; data collection continued through May 2019. Recruitment and data collection during the provision of clinical services within three community clinics that were embedded within neighborhood centers regularly accessed by the community (i.e., afterschool care centers, family and neighborhood resource programs).
Pre-assignment Details: Caregivers and children were considered enrolled in the current study. Caregivers were recruited based on their participation in a parenting intervention for their child. The Enrollment number and number of participants Started/Completed represents the number of dyads (caregiver+child). For example, 39 caregivers started treatment with their child in the CA+CFI group and 50 caregivers started treatment with their child in the CA only group.
Period: Overall Study
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Started | 39 (1. Caregivers=39, Children=39) | 50 (Caregivers=50, Children=50)
Completed | 18 (Caregivers=18, Children=18) | 20 (Caregivers=50, children=50)
Not Completed | 21 | 30
Not completed — Caregiver/child dyad dropped out before completing a full course of treatment | 21 | 30

BASELINE CHARACTERISTICS:
Population: CA + CFI group = 39 caregivers and 39 children (39 caregiver/child dyads). CA only group = 50 caregivers and 50 children (50 caregiver/child dyads)
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only | Total
Number analyzed (Participants) | 78 | 100 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: CA + CFI group = 39 caregivers and 39 children (39 caregiver/child dyads). CA only group = 50 caregivers and 50 children (50 caregiver/child dyads)
  years
    Child Age: number analyzed (Participants) | 39 | 50 | 89
    Child Age | 5.2 (1.6) | 5.03 (1.5) | 5.1 (1.6)
    Caregiver Age: number analyzed (Participants) | 39 | 50 | 89
    Caregiver Age | 35.1 (7.4) | 33.8 (70) | 34.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We only have sex data available for the child, not the caregiver. There are n=39 children in the CA+CFI group and n=50 children in the CA only group.
  Participants
    Child Sex: number analyzed (Participants) | 39 | 50 | 89
    Child Sex: Female | 11 | 17 | 28
    Child Sex: Male | 28 | 33 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total number of participants= 78 for the CA+CFI group (39 caregivers + 39 children); =100 for CA only group (50 caregivers + 50 children)
  Participants
    Child Race: number analyzed (Participants) | 39 | 50 | 89
    Child Race: American Indian or Alaska Native | 1 | 0 | 1
    Child Race: Asian | 1 | 0 | 1
    Child Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child Race: Black or African American | 11 | 8 | 19
    Child Race: White | 22 | 34 | 56
    Child Race: More than one race | 4 | 4 | 8
    Child Race: Unknown or Not Reported | 0 | 4 | 4
    Primary Caregiver Race: number analyzed (Participants) | 39 | 50 | 89
    Primary Caregiver Race: American Indian or Alaska Native | 1 | 0 | 1
    Primary Caregiver Race: Asian | 1 | 0 | 1
    Primary Caregiver Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Primary Caregiver Race: Black or African American | 12 | 9 | 21
    Primary Caregiver Race: White | 22 | 34 | 56
    Primary Caregiver Race: More than one race | 3 | 2 | 5
    Primary Caregiver Race: Unknown or Not Reported | 0 | 5 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Total number of participants= 78 for the CA+CFI group (39 caregivers + 39 children); =100 for CA only group (50 caregivers + 50 children)
  Participants
    Child Ethnicity: number analyzed (Participants) | 39 | 50 | 89
    Child Ethnicity: Hispanic/Latinx | 21 | 35 | 56
    Child Ethnicity: Haitian | 1 | 3 | 4
    Child Ethnicity: Non-Hispanic or Haitian | 17 | 12 | 29
    Primary Caregiver Ethnicity: number analyzed (Participants) | 39 | 50 | 89
    Primary Caregiver Ethnicity: Hispanic/Latinx | 20 | 36 | 56
    Primary Caregiver Ethnicity: Haitian | 2 | 2 | 4
    Primary Caregiver Ethnicity: Non-Hispanic or Haitian | 17 | 12 | 29
Income to needs ratio [Mean (Standard Deviation); unit: ratio] — Incometo-needs (INR) ratios were computed by dividing their total household income by the Federal Poverty Threshold (FPT) based on their family's size in 2018-2019. The ratio reflects household income relative to the poverty threshold, and categorized as "extreme poverty" (INR ≤ .5), "poor" (.5< INR ≤1), "low-income" (1< INR ≤2), "adequate-income" (2< INR ≤4), and "affluent" (INR > 4). Population: The income to needs ratio is reported for each caregiver/child dyad (n=89), not individually for the child and the caregiver.
  ratio
    number analyzed (Participants) | 39 | 50 | 89
    (all) | 2.2 (2.8) | 2.6 (4.01) | 2.4 (3.5)
Caregiver Education [Count of Participants; unit: Participants] — Population: Caregiver education is reported only for the caregiver (total N=89), not individually for the child and the caregiver.
  CA+CFI=39 caregivers CA only=50 caregivers
  Participants
    number analyzed (Participants) | 39 | 50 | 89
    < High School | 4 | 10 | 14
    High School/GED | 12 | 15 | 27
    Some College/AA | 8 | 9 | 17
    Bachelor's Degree | 8 | 9 | 17
    Graduate Degree | 7 | 7 | 14
Everyday Stressors Index [Mean (Standard Deviation); unit: scores on a scale] — The Everyday Stressors Index (ESI) is 20-item measure of daily stressors experienced by economically disadvantaged caregivers with young children. Items are rated on a Likert-style scale ranging from 1 = "not at all bothered" to 4 = "bothered a great deal," as well as "I don't know" = 0, and tallied with higher scores indicating greater daily stress (Scores can range from 0-80). Population: Everyday Stressors Index is reported for each caregiver/child dyad (total N=89), not individually for the child and the caregiver.
  CA+CFI = 39 caregiver/child dyad CA only = 50 caregiver/child dyad
  scores on a scale
    number analyzed (Participants) | 39 | 50 | 89
    (all) | 32.6 (6.9) | 34.7 (9.3) | 33.8 (8.4)
Eyberg Child Behavior Inventory [Mean (Standard Deviation); unit: units on a scale] — The Eyberg Child Behavior Inventory (ECBI; Eyberg & Pincus,1999) is a 36-item parent-report measure of disruptive behavior problems in children from age 2 to 18. The ECBI contains an Intensity scale that measures the frequency of disruptive behaviors . Parents rate the intensity of their child's behavior on a Likert-style scale from 1 = 'not at all frequently' to 7 = 'very frequently'. Individual Intensity Score items are summed up, with resultant scores ranging from 36 to 252. An ECBI score of 114 is the clinical cutoff for behavior problems. Population: Eyeberg Child Behavior Inventory is reported for each caregiver/child dyad (total N=89), not individually for the child and the caregiver.
  CA+CFI = 39 caregiver/child dyad CA only = 50 caregiver/child dyad
  units on a scale
    number analyzed (Participants) | 39 | 50 | 89
    (all) | 157.1 (34.2) | 149.2 (27.2) | 152.9 (30.7)

OUTCOME MEASURES:

1. Primary Outcome: CFI Clinician Questionnaire
Description: The CFI Clinician Questionnaire is a 4-item measure developed designed to assess clinical utility of the CFI. Items are rated on a 5-point Likert style scale ranging from 1='not at all' to 5='very much'. Each item has a minimum score of 1 and a max of 5. Items include the extent to which conducting the CFI influences content and quality of information obtained in the intake, realtionship with the caregiver, treatment planning, and differential diagnosis. Higher scores indicate higher levels of clinical utility of the CFI. The measure was given only to the CA + CFI condition.
  This analysis was utilized to assess for initial utility of the CFI and was mistakenly entered into the system as a primary outcome variable. This measure is not used to determine the effect of an experimental variable on participants in the study. Statistical analyses for this measure were descriptive and only examined for the experimental group.
Time Frame: Post Intake Assessment (Week 0)
Population: Descriptive analyses were conducted to assess clinical utility.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Assessment and CFI
Number analyzed (Participants) | 39
units on a scale
  Quality of Information Received | 4.2 (.59)
  Relationship with Caregiver | 4.1 (.92)
  Treatment Planning | 3.8 (.89)
  Differential Diagnosis | 3.6 (1)

2. Primary Outcome: Satisfaction With Intake Questionnaire
Description: The Satisfaction with Intake Questionnaire is a 7-item measure developed for use in the current study to assess parent and clinician satisfaction with their intake assessment. This measure assesses how well the patient/clinician felt the clinician understood the family's problems, cultural background, how their culture may influence their problem, and how much the parent trusts the clinician. Items are rated on a 5-point Likert style scale ranging from 1='not at all' to 5='very much', with higher scores representing higher satisfaction. Each item has a minimum of 1 and maximum of 5. Items were not summed.
  Two items were analyzed separately for the main outcomes: linear regressions tested condition effects on caregiver and provider satisfaction, and the extent to which the provider understood the caregivers' values or what is important to them.
Time Frame: Post Intake Assessment (Week 0)
Population: Linear regressions tested condition effects on caregiver and provider satisfaction, and the extent to which the provider understood the caregivers' values or what is important to them.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
units on a scale
  Caregiver Post-Assessment Perceptions and Satisfaction: Provider understands family values | 4.48 (.93) | 4.32 (.88)
  Caregiver Post-Assessment Perceptions and Satisfaction: Overall Satisfaction | 4.61 (.93) | 4.7 (.75)
  Provider Post-Assessment Perceptions and Satisfaction: Understands family values | 4.57 (.99) | 4.12 (.73)
  Provider Post-Assessment Perceptions and Satisfaction: Overall Satisfaction | 4.66 (.7) | 4.52 (.71)
Statistical Analysis 1: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. This linear regressions tested condition effects on caregiver perceptions of the extent to which the provider understood the caregivers' values or what is important to them; Test type: Superiority — Due to condition differences all analyses controlled for length of intake assessment (in minutes), site, caregiver race/ethnicity, daily stress, and language of assessment delivery; p = .03, Regression, Linear
Statistical Analysis 2: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed.This linear regressions tested condition effects on caregiver satisfaction with the intake; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .68, Regression, Linear
Statistical Analysis 3: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed.This linear regressions tested condition effects on provider perceptions of the extent to which the provider understood the caregivers' values or what is important to them; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .03, Regression, Linear
Statistical Analysis 4: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. This linear regressions tested condition effects on provider satisfaction with the intake; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < .05, Regression, Linear

3. Primary Outcome: CFI Fidelity Instrument
Description: The CFI Fidelity Instrument assesses fidelity to the CFI (i.e. adherence and competence) in the CA+CFI group and potential cross-condition contamination in CA condition. Independent evaluators masked to condition, study design, and study hypotheses coded recordings of all assessments.
  This analysis was utilized to assess for feasibility of the pilot study and was mistakenly entered into the system as a primary outcome variable. This measure is not used to determine the effect of an experimental variable on participants in the study. Statistical analyses for this measure were only descriptive.
Time Frame: Post Intake Assessment (Week 0)
Population: Descriptive analyses were conducted to assess clinician fidelity to the CFI and potential cross contamination given therapists delivered both conditions. The percentage was calculated by dividing the number of adherent items by number of CFI items (16 items). This was averaged to come up with the overall adherence value by group.
Measure: Mean (Standard Deviation); unit: percentage of adherence to CFI
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
percentage of adherence to CFI | 84.4 (21.5) | 4.8 (10.5)

4. Secondary Outcome: Working Alliance Inventory-Short Form Revised
Description: The WAI-Short Form Revised (WAI-SR; Hatcher & Gillaspy, 2006) is a 12-item clinician- and patient-report measure of therapeutic alliance that assesses (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Items are rated on a 5-point Likert style scale ranging from 1='never' to 5='always'. Scores on each sub scale are summed to create a total score. Total scores range from 12-60 with higher scores representing higher therapeutic alliance.
Time Frame: Post Treatment (Anticipated average: Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
score on a scale | 54.03 (8.9) | 57.06 (7.21)
Statistical Analysis 1: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. Linear regressions tested condition effects on therapeutic alliance; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .93, Regression, Linear
Statistical Analysis 2: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Tested the moderation effects of language of service reception and condition on therapeutic alliance; Test type: Superiority; p = .90, Regression, Linear

5. Secondary Outcome: Treatment Response
Description: Treatment response reflected traditional PCIT graduation criteria: caregiver skill acquisition as coded against specific criteria in both phases of treatment; and (b) child behavior problems dropped into the subclinical range.
  Families were classified as Treatment Responders in accordance with formal PCIT graduation criteria, that is: (a) caregivers demonstrated skill acquisition, as coded against specific criteria in both phases of treatment; and (b) child behavior problems dropped into the subclinical range - i.e., Eyberg Child Behavior Inventory (ECBI) falls below 114).
  Participants were coded as either treatment responders=1, or treatment non-responders=0.
Time Frame: Change from Baseline (Week 0) through post treatment (anticipated average: Week 14)
Population: Treatment response is a dichotomous variable the data presented below is probability for those variables.
Measure: Number; unit: probability treatment response
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
probability treatment response | .53 | .35
Statistical Analysis 1: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. A logistic regression tested condition effects on treatment response; Test type: Superiority — Due to condition differences all analyses controlled for length of intake assessment (in minutes), site, caregiver race/ethnicity, daily stress, and language of assessment delivery. Baseline ECBI score was included as a covariate for the treatment response analyses; p = .171, Regression, Logistic
Statistical Analysis 2: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Testes the effects of the moderation of language of service delivery and condition on treatment response; Test type: Superiority; p < .05, Regression, Logistic

6. Secondary Outcome: Engagement
Description: Engagement will be measured for each family via: (a) dichotomous coding of initial session attendance (yes=1, no=0), (b) dichotomous coding of whether they completed the first treatment module (yes=1, no=0), (c) attendance rate (number of sessions attended over number of weeks in treatment), and (d) mean weekly homework completion across treatment (Homework Compliance)
Time Frame: Change from Baseline (Week 0) through post treatment
Population: Initial session completion, and completion of first treatment modules are dichotomous variables the data presented below is probability for those variables.
Measure: Number; unit: probability of engagement
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
probability of engagement
  Session Attendance | .65 | .57
  Homework Completion | .49 | .46
  Initial Session Attendance | .95 | .91
  Completion of first treatment modules | .75 | .35
Statistical Analysis 1: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. Linear regressions tested condition effects on session attendance; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .38, Regression, Linear
Statistical Analysis 2: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Analyses tested the moderation of language of service delivery and condition on session attendance; Test type: Superiority; p = .01, Regression, Linear
Statistical Analysis 3: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. linear regressions tested condition effects on homework completion. Due to condition differences all analyses controlled for length of intake assessment (in minutes), site, caregiver race/ethnicity, daily stress, and language of assessment delivery; Test type: Superiority; p = .56, Regression, Linear
Statistical Analysis 4: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Analyses tested the moderation effect of language of service delivery and condition on homework completion; Test type: Superiority; p < .01, Regression, Linear
Statistical Analysis 5: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. Logistic regressions tested condition effects on initial session attendance. Due to condition differences all analyses controlled for length of intake assessment (in minutes), site, caregiver race/ethnicity, daily stress, and language of assessment delivery; Test type: Superiority; p = .40, Regression, Logistic
Statistical Analysis 6: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Analyses tested the moderation of language of service delivery and condition on initial session attendance; Test type: Superiority; p = .01, Regression, Logistic
Statistical Analysis 7: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. A Logistic regression tested condition effects on completion of first treatment module. Due to condition differences all analyses controlled for length of intake assessment (in minutes), site, caregiver race/ethnicity, daily stress, and language of assessment delivery; Test type: Superiority; p = .03, Regression, Logistic
Statistical Analysis 8: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; Analyses tested the moderation of language of service delivery and condition on completion of first treatment module; Test type: Superiority; p = .03, Regression, Logistic

7. Secondary Outcome: Therapy Attitudes Inventory
Description: The Therapy Attitudes Inventory (TAI; Brestan et al., 2000) is a 10-item parent-report of satisfaction with treatment including change in child behavior problems and parenting skills on a likert style scale from 1="nothing"-5="very many useful techniques". Items are summed to create a total score. Minimum value is 10 and maximum value is 50. Higher scores represent higher satisfaction with treatment.
Time Frame: Post Treatment (anticipated average: Week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
score on a scale | 48.490 (3.63) | 48.581 (2.58)
Statistical Analysis 1: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. linear regressions tested condition effects on treatment satisfaction; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .854, Regression, Linear

8. Secondary Outcome: Eyberg Child Behavior Inventory
Description: The Eyberg Child Behavior Inventory (ECBI; Eyberg & Pincus, 1999) is a 36-item parent-report measure of disruptive behavior problems in children as young as 2 years that has shown strong psychometrics. The intensity score is summed to form a total score and ranges from 36 to 252 with higher numbers representing more severe behavior problems.
  The difference in ECBI score between baseline and treatment completion was measured.
Time Frame: Change from Baseline (Week 0) through post treatment (anticipated average: Week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
units on a scale | 46.35 (42.67) | 51.737 (39.47)
Statistical Analysis 1: Comparison: Clinical Assessment and CFI vs Clinical Assessment Only; A power analysis assuming an alpha level = 0.05, beta = 0.2, and power = 0.8, identified a sample ≥82 participants was needed to identify small-to-medium effects (i.e., OR~2.5).Intent-to-treat analyses were employed. linear regressions tested change in ECBI score from baseline to post treatment; Test type: Superiority; p = .319, Regression, Linear

9. Secondary Outcome: Everyday Stressors Index
Description: The Everyday Stressors Index (ESI Hall, 1983) is a 20-item measure that assesses daily stressors experienced by economically disadvantaged parents with young children. Items are rated on a Likert-style scale ranging from 1='not at bothered' to 4='bothered a great deal' with higher scores indicating higher levels of stress. The minimum value=20, and maximum value=80
  This is a single time point assessment and is therefore not an outcome variable. There was an error when registering in clinical trials.
Time Frame: Post Intake Assessment (Week 0)
Population: This is a single time point assessment and is therefore not an outcome variable. There was an error when registering in clinical trials. Only baseline descriptive data is provided.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
score on a scale | 32.6 (6.9) | 34.7 (9.3)

10. Secondary Outcome: Multigroup Ethnic Identity Measure- Revised
Description: The Multigroup Ethnic Identity Measure- Revised (MEIM-R; Phinney & Ong, 2007) is a 6-item measure that assesses exploration of and commitment to one's ethnic group. Items are rated on a 5-point Likert-style scale from 1='strongly disagree' to 6='strongly agree', with higher scores indicating stronger ethnic identity.
  This is a single time point assessment and is therefore not an outcome variable. There was an error when registering in clinical trials.
Time Frame: Post Intake Assessment (Week 0)
Population: This is a single time point assessment and is therefore not an outcome variable. There was an error when registering in clinical trials.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
score on a scale | 2.729 (1.667) | 2.778 (.838)

11. Secondary Outcome: Parental Attitudes Toward Psychological Services Inventory
Description: Two subscales of the Parental Attitudes Toward Psychological Services Inventory (PATPSI; Turner, 2012) will be administered: help seeking attitudes scale (8 items) and the stigmatization scale (8 items) comprising 16 items total. The PATPSI assesses caregivers' attitudes toward outpatient mental health services. Items are rated on a 5-point Likert-style scale from 0='strongly disagree' to 5='strongly agree'.
  Item responses are summed to form a stigma total scale (minimum value=0 and maximum value=40) and a help seeking total scale (minimum value=0 and maximum value=40) with higher scores representing more mental health related stigma and more positive attitudes toward mental health services.
  This is a single time point assessment and is therefore not an outcome variable. There was an error when registering in clinical trials.
Time Frame: Post Intake Assessment (Week 0)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
score on a scale
  Stigma Subscale | 5.847 (5.19) | 6.172 (5.57)
  Help Seeking Subscale | 6.384 (5.718) | 6.970 (6.097)

12. Secondary Outcome: Everyday Discrimination Scale
Description: The Everyday Discrimination Scale (EDS; Williams et al., 1997) is a 9-item measure that assesses aspects of interpersonal discrimination or unfair treatment in their day-to-day life. Items are rated on a Likert-style scale ranging from 0='never' to 5='almost every day', with higher scores indicating more experiences of discrimination. The minimum score is 0 and maximum score is 45. Scores were averaged to create a mean discrimination score which could range from 0 to 5.
  This is a single time point assessment and is therefore not an outcome variable. There was an error when registering in clinical trials.
Time Frame: Post Intake Assessment (Week 0)
Population: This is a single time point assessment and is therefore not an outcome variable. There was an error when registering in clinical trials. Online baseline data is provided.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
Number analyzed (Participants) | 39 | 50
score on a scale | .806 (.746) | .658 (.627)

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Arm/Group | Clinical Assessment and CFI | Clinical Assessment Only
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/50
Other Adverse Events (participants affected / at risk) | 0/39 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT03499600/Prot_SAP_000.pdf